CLINICAL TRIAL: NCT00002638
Title: HIGH-DOSE CHEMOTHERAPY FOLLOWED BY AUTOLOGOUS PERIPHERAL BLOOD STEM CELL TRANSPLANTATION FOR CHILDREN WITH RELAPSED ACUTE LYMPHOCYTIC LEUKEMIA
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Children With Relapsed Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: UNMC-06695; CDR0000064114 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0639
Record Dates: First submitted 1999-11-01; First posted 2003-09-18 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2002-09

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; sargramostim; Carmustine; Cyclophosphamide; Cytarabine; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation in treating children who have relapsed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of autologous peripheral blood stem cell (PBSC) transplantation for marrow reconstitution after high-dose carmustine, cytarabine, etoposide, and cyclophosphamide in children with relapsed acute lymphocytic leukemia.
* Determine the dose effect of autologous PBSC on engraftment in this patient population.

OUTLINE: Patients receive chemotherapy mobilization comprising cytarabine IV every 12 hours on days 1-5. When blood counts recover, autologous peripheral blood stem cells (PBSC) are harvested and selected for mononuclear cells, granulocyte-macrophage colony-forming units, and CD34+ cells.

Patients receive preparative regimen comprising carmustine IV on days -8 and -3, cytarabine IV every 12 hours and etoposide IV every 12 hours on days -7 to -4, and cyclophosphamide IV on days -2 and -1. PBSC are reinfused on day 0. Patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) beginning after PBSC transplantation. Male patients undergo radiotherapy to the testes before transplantation. Patients with a history of CNS leukemia undergo craniospinal irradiation before transplantation.

Patients are followed at 100 days, 6 months, and 1 year.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia

  * Pathologic evidence of relapse in marrow, CNS, or testes
  * In second or later complete remission
* Ineligible for allogeneic transplantation:

  * No suitable allogeneic donor (sibling or family donor or unrelated donor with no more than 1 HLA-A or -B antigen mismatch and HLA-DR identical) OR
  * Ineligible for preparative regimen including total-body irradiation
* Peripheral blood stem cell collection feasible:

  * Patient size generally at least 8 kg
  * Able to place central venous catheter
  * Patient cooperative

PATIENT CHARACTERISTICS:

Age:

* 1 to 19

Performance status:

* Not moribund

Life expectancy:

* No severe limits from disease other than leukemia

Hepatic:

* Bilirubin no greater than 3 times normal for age
* AST and/or GGT no greater than 3 times normal for age
* No evidence of hepatic synthetic dysfunction

Renal:

* GFR at least 50% of normal based on Glofil study or 12-hour creatinine clearance

Cardiovascular:

* Cardiac contractility normal on echocardiogram

Pulmonary:

* FVC and FEV_1 with or without DLCO at least 50% predicted

Other:

* No significant active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1995-03; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Gordon, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States